CLINICAL TRIAL: NCT02435342
Title: A 4 Week Study of the Safety, Tolerability, and Pharmacodynamics of ShK-186 in Active Plaque Psoriasis
Brief Title: A 4 Week Study of the Safety, Tolerability, and Pharmacodynamics of ShK-186 (Dalazatide) in Active Plaque Psoriasis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kineta Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 186-03
Record Dates: First submitted 2015-04-15; First posted 2015-05-06 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-05

CONDITIONS: Plaque Psoriasis
Keywords: ShK-186; dalazatide; psoriasis; Kv1.3,; autoimmune
MeSH Terms: conditions — Psoriasis | interventions — Shk-186 peptide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 30ug dalazatide (Experimental): 12 subjects, 10 given active agent and 2 given placebo by subcutaneous injection twice weekly for 4 weeks.
  Interventions: Drug: dalazatide; Drug: placebo
- 60ug dalazatide (Experimental): 12 subjects, 10 given active agent and 2 given placebo by subcutaneous injection twice weekly for 4 weeks.
  Interventions: Drug: dalazatide; Drug: placebo

INTERVENTIONS:
Drug: dalazatide — Subcutaneous injection twice per week for a total of 9 doses, followed by four weeks of follow-up.
  Other Names: ShK-186
Drug: placebo — placebo, Subcutaneous injection twice per week for a total of 9 doses

SUMMARY:
The primary purpose of this study is to examine safety outcomes in active plaque psoriasis patients after systemic administration of dalazatide. Clinical outcome measures will also be assessed.

DETAILED DESCRIPTION:
The primary purpose of this study is to examine safety outcomes in active plaque psoriasis patients after systemic administration of dalazatide. Clinical outcome measures will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male and female subjects, ages 18-65;
2. Active plaque psoriasis with ≥3% BSA involved;
3. An adequate number of vulgar psoriatic plaques of at least 2 cm X 2 cm with Target Lesion Investigator Global Assessment scores >3, that are not located on the face, scalp, groin, genitals, folds, palms or soles
4. Weight of 50 - 100 kg;
5. Non-child bearing potential or willingness to use adequate contraception in order to prevent pregnancy from the screening visit until 60 days after the follow-up visit.
6. Subject will be evaluated for latent TB infection.
7. Able to communicate and able to provide valid, written informed consent;

Exclusion Criteria:

The following will exclude potential subjects from the study:

1. Erythrodermic, predominantly guttate, exclusively palmar/plantar, or generalized pustular psoriasis;
2. Current drug-induced or aggravated psoriasis (e.g., a new onset of psoriasis or an exacerbation of psoriasis from beta-blockers, calcium-channel blockers, or lithium carbonate);
3. Use of the following concurrent systemic medications: corticosteroids, retinoids, cyclosporine, methotrexate, or biologic agents.
4. Use of concurrent topical medications (must be discontinued at least 2 weeks prior to baseline);
5. UVA or UVB therapy within 4 weeks of baseline;
6. The presence of uncontrolled hypertension, uncontrolled diabetes, clinically significant cardiovascular disease, asthma or reduced pulmonary capacity, or a history of seizure or other neurologic disorder;
7. Presence or history of pre-existing paresthesia or neuropathy;
8. Abnormalities on neurological exam at screening or baseline;
9. Clinically significant ECG abnormalities, in the opinion of the Investigator;
10. History of any cancer requiring systemic chemotherapy or radiation;
11. The presence of acute infection or history of acute infection as judged by the Investigator within 7 days of baseline;
12. The presence of clinically significant laboratory abnormalities;
13. A positive hepatitis screen (Hepatitis BsAg or anti-HCV) or positive Human Immunodeficiency Virus (HIV) antibody test ;
14. History of treated or untreated TB
15. Any history of anaphylaxis that is important in the view of the Investigator;
16. Participation in another clinical trial with receipt of an investigational product within 90 days of baseline (or 5 half-lives of the previous drug, whichever is longer);
17. History of alcohol abuse that is important in the view of the Investigator;
18. Positive drug screen for amphetamines, barbituates, benzodiazepines, cocaine, cannabis, methamphetamine, methylenedioxymethanphetamine, opiates or phencyclidine
19. Inadequate venous access that would interfere with obtaining blood samples;
20. Positive pregnancy test at screening or at baseline or current lactation (female subjects only);
21. Inability or unwillingness to comply with study restrictions, return for follow up appointments, or other considerations, in the opinion of the Investigator, which would make the candidate unsuitable for study participation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-10; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Subjects with adverse events | From randomization through Day 57 (12 timepoints)

SECONDARY OUTCOMES:
Target lesion assessment | From randomization to Day 57 (4 timepoints)
  Target lesion evaluated for erythema, induration, and scaling.
Psoriasis Area Severity Index (PASI) score | From randomization to Day 57 (4 timepoints)
Patient and Investigator Global Assessment of Psoriasis | From randomization to Day 57 (4 timepoints)
Psoriasis Disability Index (PDI) | From randomization to Day 57 (4 timepoints)
Skin biomarker assessments | From randomaization to Day 32 (2 timepoints)
  Skin biopsy from psoriatic lesion collected for analysis of gene expression via qPCR and immune cell infiltration via histology and immunohistochemistry analysis.
Blood biomarker assessments | From randomizatoin to Day 57 (5 timepoints)
  Blood collected for analysis of gene and protein expression as well as immunophenotyping of T cell subsets.
Dermatology Quality of Life Questionnaire (DLQI) | From randomization to Day 57 (4 timepoints)
Presence of specific anti-drug antibodies to dalazatide | From randomization to Day 57 (three timepoints)
  Serum evaluated for specific anti-drug antibody using ELISA-based immunoassay.
Subjects with changes in vital signs | From randomization to Day 57 (12 timepoints)
  Vital signs include temperature, respiratory rate, supine blood pressure and pulse.
Subjects with changes in symptom-directed physical examinations | From randomization to day 5 (12 timepoints)

OTHER OUTCOMES:
Area under the plasma concentration versus time curve of dalazatide (AUC) | 5 minutes pose dose, 15 minutes post dose, 30 minutes post dose, 1 hour post dose, 2 hours post dose, 4 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Shawn Iadonato, PhD, Study Director — Kineta Inc.
Locations (1):
- Innovaderm Research, Inc, Montreal, Quebec, Canada